CLINICAL TRIAL: NCT03615105
Title: Allogeneic Hematopoietic Cell Transplantation Using α/β+ T-lymphocyte Depleted Grafts From HLA Mismatched Donors
Brief Title: Donor Stem Cell Transplantation Using α/β+ T-lymphocyte Depleted Grafts From HLA Mismatched Donors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-224
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-03

CONDITIONS: Acute Lymphoid Leukemia (ALL); Acute Myeloid Leukemia (AML); Chronic Myeloid Leukemia (CML); Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: Allogeneic Hematopoietic Cell Transplantation; α/β+ T-lymphocyte; 18-224
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Thiotepa; Cyclophosphamide; Busulfan; fludarabine; Melphalan; Clofarabine; Rituximab

STUDY DESIGN:
Intervention Model Description: Participants will receive one of three myeloablative conditioning regimens followed by a Alpha/beta+ T-cell depleted peripheral blood stem cell product and short course tacrolimus. Donors are HLA mismatched unrelated adults or haploidentical family members.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Radiation, Thiotepa & Cyclophosphamide (Experimental)
  Interventions: Radiation: Hyperfractionated total body irradiation; Drug: Thiotepa; Drug: Cyclophosphamide; Procedure: HPC(A) stem cell allograft; Drug: Rituximab; Device: Rabbit antithymocyte globulin
- Busulfan, Fludarabine & Melphalan (Experimental)
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: Melphalan; Procedure: HPC(A) stem cell allograft; Drug: Rituximab; Device: Rabbit antithymocyte globulin
- Clofarabine, Thiotepa & Melphalan (Experimental)
  Interventions: Drug: Thiotepa; Drug: Melphalan; Drug: Clofarabine; Procedure: HPC(A) stem cell allograft; Drug: Rituximab; Device: Rabbit antithymocyte globulin

INTERVENTIONS:
Radiation: Hyperfractionated total body irradiation — Hyperfractionated TBI is administered by a linear accelerator at a dose rate of <20 cGy/minute. Doses of 125 cGy/fraction are administered at a minimum interval of 4 hours between fractions, three times/day for a total of 11 or 12 doses (1,375 or 1,500 cGy) over 4 days (days -9 through -6).
  Arms: Radiation, Thiotepa & Cyclophosphamide
Drug: Thiotepa — Thiotepa 5 mg/kg IV
  Arms: Clofarabine, Thiotepa & Melphalan; Radiation, Thiotepa & Cyclophosphamide
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg IV
  Arms: Radiation, Thiotepa & Cyclophosphamide
Drug: Busulfan — Busulfan (adult/ped dose)
  Arms: Busulfan, Fludarabine & Melphalan
Drug: Fludarabine — Fludarabine 25 mg/m2 IV
  Arms: Busulfan, Fludarabine & Melphalan
Drug: Melphalan — Melphalan 70 mg/m2 IV
  Arms: Busulfan, Fludarabine & Melphalan; Clofarabine, Thiotepa & Melphalan
Drug: Clofarabine — Clofarabine 20-30 mg/m2 IV
  Arms: Clofarabine, Thiotepa & Melphalan
Procedure: HPC(A) stem cell allograft — All patients will receive anti-thymocyte globulin based conditioning followed by a G-CSF mobilized, peripheral blood hematopoietic progenitor cell HPC(A) product depleted of TCR-α/β+ Tlymphocytes using the CliniMACS system.
Drug: Rituximab — Rituximab 200 mg IV flat dose
Device: Rabbit antithymocyte globulin — Rabbit antithymocyte globulin dosing per nomogram. This dynamic nomogram is based on absolute lymphocyte count at the start of conditioning and can result in either 2 or 3 day ATG administration. If a patient requires 2 day administration the subjequent chemotherapies may be moved forward by one day at the treating physician's discretion.

SUMMARY:
This study is being done to learn whether a new method to prevent rejection between the donor immune system and the patient's body is effective.

ELIGIBILITY:
Subject Inclusion Criteria:

* Patients with any of the following hematologic malignancies who are considered to be eligible for allogeneic transplantation:

  * Acute lymphoid leukemia (ALL) in first complete remission (CR1) with high risk for relapse including:

    * Detectable minimal residual disease by either multicolor flow cytometry or by genomic assay after initial induction therapy
    * t(9;22) or detected BCR-ABL1 translocation by genomic methodologies
    * BCR-ABL1-Like B-ALL [23] including mutations of IKZF1 or CRLF2
    * Translocations or mutations involving 11q23 (MLL) gene.
    * Hypodiploid karyotype
    * Deletion of 9p
    * Loss of 17p or TP53 mutation
    * T-lymphocyte lineage antigen expression (T-ALL)
    * Prior CNS or other extramedullary involvement
    * WBC count ≥ 100,000 cells/μL at diagnosis
    * Acute biphenotypic or bilineal leukemia in CR1
  * Acute myeloid leukemia (AML) in CR1 with

    * Detectable minimal residual disease (MRD) by either multicolor flow cytometry or by genomic assay after initial induction therapy
    * In the absence of MRD any intermediate or high risk features according to the European LeukemiaNet 2017 guidelines indlucing:
* Mutated FL T3-ITD or FL T3-TKD
* Cytogenetic abnormalities not classified as favorable
* Cytogenetic abnormalities associated with myelodysplastic syndrome including abnormalities of chromosome 5, 7, or 17p
* Complex karyotype or monosomal karyotype
* t(9;11)(p21.1;q23.3); MLL-KMT2A or other rearrangements of KMT2A
* t(9;11); BCR-ABL1
* Inversions or translocations of chromosome 3
* T(6;9)(p23;q34.1); DEK-NUP214
* Somatic mutation of RUNX1, ASX1 or TP53

  * Extramedullary involvement
  * WBC count ≥100,000 cells/μL at diagnosis

    * Relapsed acute leukemia with ≤ 5% blasts in the bone marrow prior to transplantation (i.e. CR2 or greater).
    * Myelodysplastic syndrome, myeloproliferative neoplasms, or MDS/MPN overlap syndrome with ≤ 10% blasts and at least one of the following:
  * Revised International Prognostic Scoring System risk score of INT, HIGH, or VERY HIGH at the time of transplant evaluation.
  * Life-threatening cytopenias
  * Karyotype or genomic changes that indicate high risk for progression to acute myelogenous leukemia, including abnormalities of chromosome 7 or 3, mutations of TP53, or complex or monosomal karyotype.
  * Therapy related disease or disease evolving from other malignant processes.

    * Chronic myelomonocytic leukemia (CMML) with ≤ 10% blasts prior to transplantation.
    * Chronic myeloid leukemia (CML) meeting one of the following criteria:
  * Failed or are intolerant to BCR-ABL tyrosine kinase inhibitors.
  * CML with BCR-ABL mutation consistent with poor response to tyrosine kinase inhibition (e.g. T351I mutation).
  * CML with accelerated or blast phase with <10% blasts after therapy.

    * Chronic lymphocytic leukemia (CLL) with high risk disease as defined by the EBMT consensus criteria
    * Hodgkin lymphoma meeting both of the following criteria:
  * Responding to therapy prior to enrollment
  * Relapse after autologous bone marrow transplant or are ineligible for autologous bone marrow transplant.

    °Non-Hodgkin lymphoma meeting both of the following criteria:
  * Responding to therapy prior to enrollment.
  * Relapse after prior autologous bone marrow transplant or are ineligible for autologous bone marrow transplant.
  * Patients aged from birth through 65 years old are eligible.
  * Patients must have Karnofsky/Lanksy performance status ≥70%.
  * Cardiac left ventricular ejection fraction ≥50% at rest.
  * Serum bilirubin ≤ 2 mg/dL. Patients with Gilbert's disease or ongoing hemolytic anemia are acceptable if the direct bilirubin is ≤ 2 mg/dL.
  * AST and ALT ≤ 2.5 x ULN unless thought to be disease related
  * Estimated or measured creatinine clearance > 50 mL/min/1.73 m^2 body surface area.
  * Adult patients and pediatric patients capable of performing pulmonary function studies must have hemoglobin adjusted pulmonary DLCO ≥50% of predicted.

Subject Exclusion Criteria:

* Persons with a HLA matched sibling donor or a 8/8 allele level HLA-matched unrelated donor.
* Female patients who are pregnant or breast-feeding.
* Persons with an infection that is not responding to antimicrobial therapy.
* Persons who are seropositive for HIV.
* Persons with active/detectable central nervous system malignancy.
* Persons who do not meet the age and organ function criteria specified above.
* Presence of psychiatric or neurologic disease, or lack of social support that limits the patient's ability to comply with the treatment protocol including supportive care, followup, and research tests.
* Prior allogeneic hematopoietic cell transplantation are ineligible.
* Patients with history of other malignancy within 5 years of study therapy are ineligible with the following exceptions: Low grade prostate cancer (Gleason's ≤6) treated with curative intent, breast ductal carcinoma in situ treated with curative intent, or nonmelanomatous skin carcinomas.

Donor Inclusion and Exclusion Criteria:

* Partially HLA-matched unrelated volunteers (allele level matched at 6-7 of 8 HLA loci: -A, -B, -C, and -DRB1) are eligible.
* Related, haploidentical donors are eligible.
* Able to provide informed consent to the donation process
* Meet standard criteria for donor collection as defined by the National Marrow Donor Program Guidelines.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shaffer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation, Thiotepa & Cyclophosphamide | Busulfan, Fludarabine & Melphalan | Clofarabine, Thiotepa & Melphalan
Started | 3 | 5 | 1
Completed | 2 | 3 | 1
Not Completed | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Death | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation, Thiotepa & Cyclophosphamide | Busulfan, Fludarabine & Melphalan | Clofarabine, Thiotepa & Melphalan | Total
Number analyzed (Participants) | 3 | 5 | 1 | 9
Age, Continuous [Mean (Full Range); unit: years] | 20 [18 to 22] | 31 [13 to 63] | 23 [23 to 23] | 26 [13 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 0 | 6
  Male | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 0 | 3 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 0 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: the Number of Incidences of Grade 3-4 Acute GVHD
Description: The intervention will be considered unpromising if the rate of GVHD is greater than 40% and promising if the rate is 20% or less. Number of participants with and without SAE will be evaluated.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation, Thiotepa & Cyclophosphamide | Busulfan, Fludarabine & Melphalan | Clofarabine, Thiotepa & Melphalan
Number analyzed (Participants) | 3 | 5 | 1
Participants
  Number of participants with SAE | 2 | 3 | 1
  Number of participants without SAE | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Radiation, Thiotepa & Cyclophosphamide | Busulfan, Fludarabine & Melphalan | Clofarabine, Thiotepa & Melphalan
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/5 | 1/1
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/5 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation, Thiotepa & Cyclophosphamide (N=3) | Busulfan, Fludarabine & Melphalan (N=5) | Clofarabine, Thiotepa & Melphalan (N=1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Gastrointestinal disorders, other (Gastrointestinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Infection and infestations, other (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation, Thiotepa & Cyclophosphamide (N=3) | Busulfan, Fludarabine & Melphalan (N=5) | Clofarabine, Thiotepa & Melphalan (N=1)
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 5 | 1
Serum amylase increased (Investigations) | 0 | 1 | 0
White blood cell decreased (Investigations) | 3 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03615105/Prot_SAP_000.pdf